CLINICAL TRIAL: NCT00249496
Title: Therapeutic Workplace Maintenance Study
Brief Title: Employment-based Reinforcement to Motivate Drug Abstinence in the Treatment of Drug Addiction. - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 2093; R01DA013107 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Use; Drug Use; Risk Behavior; Sexual Behavior
Keywords: cocaine; opioids; contingency management; sexual risk; HIV
MeSH Terms: conditions — Alcohol Drinking; Risk-Taking; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Employment Only (Active Comparator): Employment Only participants will be offered employment for one year, but these participants will not have to provide drug-free urine samples to work.
  Interventions: Behavioral: Employment Only
- Contingency Management (Experimental): Participants in the Contingency Management group will be employed for one year in a Therapeutic Workplace business and will have to provide drug-free urine samples to work and earn salary.
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Participants in the Contingency Management group will be employed for one year in a Therapeutic Workplace business and will have to provide drug-free urine samples to work and earn salary.
  Arms: Contingency Management
Behavioral: Employment Only — Employment Only participants will be offered employment for one year, but these participants will not have to provide drug-free urine samples to work.
  Arms: Employment Only

SUMMARY:
This application is a competing continuation of a grant in which we developed and pilot tested a computerized Therapeutic Workplace designed to train and employ adults as data entry operators. A randomized trial is planned over 5 years to investigate the Therapeutic Workplace business as a maintenance intervention to sustain long-term abstinence and employment. Welfare recipients in methadone treatment, actively using cocaine, and at risk for contracting or spreading HIV infection will participate in an initial Therapeutic Workplace training phase. Participants who become abstinent and skilled will be randomly assigned to an Abstinence & Employment, or an Employment Only group. Participants in the Abstinence & Employment group will be employed for one year in a Therapeutic Workplace business and will have to provide drug-free urine samples to work and earn salary. Employment Only participants will be offered employment for one year, but these participants will not have to provide drug-free urine samples to work. This study will provide a rigorous evaluation of the efficacy of the Therapeutic Workplace business as a long-term treatment of cocaine addiction and unemployment; determine the benefits of requiring daily evidence of abstinence to work; and provide information on the extent to which a Therapeutic Workplace business can become self-sustaining. This research could provide firm scientific foundation for the dissemination of Therapeutic Workplace businesses in the long-term treatment of cocaine addiction and unemployment. The main hypothesis being tested is that cocaine abstinence will be reliably maintained during the yearlong intervention evaluation period only in the group exposed to the explicit abstinence maintenance intervention. We expect that cocaine abstinence in the Abstinence and Employment group will be significantly greater than cocaine abstinence in the Employment Only group.

DETAILED DESCRIPTION:
STUDY PARTICIPANTS This study was approved by the Western Institutional Review Board. Participants were recruited in methadone clinics throughout Baltimore. Recruitment began in October 2003, and the study was completed in August 2007. Of the 251 individuals assessed for eligibility, 128 met these criteria and were invited to participate in the study.

SETTING The study was conducted at the Center for Learning and Health, Johns Hopkins School of Medicine, Baltimore, MD. The workplace included a sign-in station, a urinalysis laboratory, and three workrooms. The workrooms contained 47 computer workstations.

PRE-RANDOMIZATION PROCEDURES Intake Assessment At intake, participants signed informed consent and completed an interview. Urine samples were collected and tested for cocaine, opiates, benzodiazepines, methadone, and amphetamines. A questionnaire was administered to assess participants' capacity to operate a keyboard. The Composite International Diagnostic Interview (CIDI), 2nd ed. was administered to assess drug dependence. Other assessment tools included the Addiction Severity Index - Lite (ASI-Lite), the Risk Assessment Battery (RAB), the Wide Range Achievement Test (WRAT-3), and a reading assessment. Participants were paid $30 in vouchers for completing the interview.

Workroom and Urinalysis Procedures Eligible participants were enrolled in phase 1 and could work in the workplace from 10 AM-12 PM and 1 PM-3 PM every weekday for 6 months. During this phase, participants worked on computerized training programs designed to teach them to become data entry operators. On Monday, Wednesday and Friday, participants provided a urine sample under observation. Breath samples were tested for alcohol. Urine samples were tested for opiates and cocaine and participants received graphs showing current and prior drug test results. Participants earned a base pay of $8.00 per hour in vouchers. Additionally, participants could earn approximately $2.00 per hour in vouchers in productivity pay for working on training programs. Earnings accumulated in the participant's account until exchanged for a gift card or other approved goods and services.

Initially, participants could attend the workplace independent of their urinalysis results. This "workplace induction" continued for at least 4 weeks and until the participant worked for at least 5 min on 15 workdays. After workplace induction, participants were required to provide evidence of cocaine abstinence to work and to maintain maximum pay. Specifically, participants gained access to their workrooms if urinary benzoylecgonine concentration was <300 ng/mL or at least 20% lower per day since the last sample submitted. Participants who provided a cocaine-positive urine sample could not work until they provided a new sample that met the criteria. Upon return to work, the rate of base pay was reduced to $1.00 per hour. Base pay was then increased by $1.00 per hour every day that a participant provided a sample that met the criteria and worked at least 5 minutes until reaching $8.00 per hour. Missing samples were treated as positive. After a participant provided cocaine-negative samples for three consecutive weeks, the abstinence contingency was extended to opiates (ie, urinary benzoylecgonine and morphine concentrations of <300 ng/mL, or decreases in benzoylecgonine and morphine concentrations by at least 20% per day since the last sample submitted). After providing cocaine- and opiate-negative samples for three consecutive weeks the contingency was expanded to include alcohol if the participant had provided alcohol positive (≥0.003 ng/L) samples during the opiate and cocaine contingency period. This stepped contingency program is described in detail elsewhere.

The training programs were designed for individuals with no typing skills. The programs were divided into small steps. Participants practiced steps in one-minute intervals until meeting mastery criteria for the step. Participants earned $0.03 per 20 correct characters typed, and lost $0.01 per 2 incorrect characters typed. Additional productivity pay ranging from $0.25 to $2.00 was provided for achieving step mastery. Participants who finished the typing program proceeded to a data entry training program, which included similar productivity pay contingencies. A detailed report of the results of phase 1 is provided elsewhere.

RANDOMIZATION Eligibility for phase 2 was assessed at the end of the fifth month of phase 1. Participants who attended the workplace on at least 50% of possible days and provided urine samples that met the reinforcement criteria on at least 80% of the collection opportunities during the four weeks prior to assessment, and who attained minimal typing proficiency qualified to participate in phase 2. Individuals not meeting criteria at the end of the fifth month who were still attending the workplace at least occasionally were reevaluated in the sixth month. This reevaluation occurred for seven participants, all of whom were admitted to phase 2 of the study. After meeting phase 2 eligibility criteria, participants were randomly assigned to employment only (n = 24) or abstinence-contingent employment (n = 27), and hired as employees of the nonprofit data entry business for one year. One eligible person declined to participate in phase 2 due to fears of losing social security benefits due to employment, and another was assigned to a discontinued study group (see below). The two groups did not differ significantly on any demographic measure assessed at intake. The phase 2 participants' mean age was 43 years, 77% were female, 88% were black, and 98% were living in poverty.

All stratification and randomization procedures were computerized and carried out by a data coordinator who did not have contact with participants. Participants were stratified according to whether 50% or more of the urine samples collected during the first four weeks of the induction period were positive for opiates; whether 75% or more of these samples were positive for cocaine; and whether they achieved an exceptionally high level of tying proficiency. Personnel who conducted monthly assessments were blind to group assignment.

POST-RANDOMIZATION PROCEDURES Phase 2 Assessments An interview was conducted immediately prior to randomization that included drug testing, the ASI-Lite, the RAB, the Vocational Educational Assessment (VEA, for assessing attitudes about work and employment history), and the Treatment Services Review (TSR, for assessing the use of professional services), and questionnaires covering adverse events and workplace satisfaction. These assessments were repeated every 30 days, except for the RAB, which was only conducted during the 6th and 12th months.

Phase 2 Employment Procedures Upon enrollment in phase 2, participants began employment as data entry operators in Hopkins Data Services.40 While employed by Hopkins Data Services, participants could work from 9 AM to 4 PM, with 1 hour for lunch. Participants earned an hourly wage slightly higher than or equal to the legal minimum (originally $5.25 per hour, but increased to $6.15 per hour when the minimum wage in Maryland increased) and pay for productivity. Contingencies for productivity pay were programmed such that participants would earn approximately $4.00 per hour in productivity pay for normative performance. Participants received regular bi-weekly paychecks instead of vouchers. Although prior employees of Hopkins Data Services performed data entry jobs for paying customers,40 given the nature of the control group (ie, no contingencies on drug abstinence), participants in this study performed data entry jobs in which they entered data batches from completed orders.

Study Groups Participants assigned to the abstinence-contingent employment group were required to provide drug negative urine samples to access the workrooms on mandatory collection days . Initially, all Mondays, Wednesdays, and Fridays were mandatory days. If a participant in this group provided a positive sample or failed to provide a sample on a mandatory day, then the participant was denied access to the workplace on that day, and until the participant provided a sample that met the criteria. In addition, participants whose urine sample did not meet the criteria were given a reset in productivity pay from $4.00 per hour to $1.00 per hour. After a reset, a participant's productivity pay increased by $1.00 per hour per day that the participant worked for a minimum of five minutes, until the standard rate of approximately $4.00 per hour was reinstated.

Participants in the abstinence-contingent employment group who provided urine samples that met the criteria on 30 consecutive calendar days were placed on a random mandatory urine testing schedule. Initially, a schedule was established in which an average of one out of every two Mondays, Wednesdays, and Fridays were designated as mandatory collection and testing days. After every 30 days in which all mandatory samples met the abstinence criteria the average was further reduced by one, until an average of one out of every six Mondays, Wednesdays, and Fridays were randomly designated as mandatory days. Participants could call the workplace to inquire whether that day's urine sample collection was mandatory. If a participant provided a positive sample on a mandatory day or missed a mandatory sample then routine mandatory testing was reinstated and the schedule-thinning process repeated from the beginning. Participants were informed of schedule changes by the workplace manager and given a written notice describing the change. Participants received urinalysis feedback graphs similar to phase 1, however, only the results of mandatory tests were displayed on the graph.

Participants assigned to the employment only group were required to provide urine samples, but were permitted to work independent of the results of urinalysis. Rate of pay was also unaffected by the urinalysis results. In order to equate the urinalysis feedback across groups, employment only participants were placed on a thinning schedule of feedback in which the progressive thinning occurred every 30 days, independent of the participant's urinalysis results. Urine samples from participants in both groups were collected for data purposes every Monday, Wednesday, and Friday that a participant attended the workplace, although participants were only given feedback about the urinalysis results on selected days.

ELIGIBILITY:
Inclusion Criteria:

* Applicants in methadone treatment may be eligible to participate in Phase 1 of the study.
* Applicants will be blind to the full details of the eligibility criteria.
* Unemployed
* Provided a urine sample at intake with a detectable concentration of cocaine metabolite or provided a cocaine positive sample during regular urinalysis testing at a methadone maintenance program
* Met DSM-IV criteria for cocaine dependence
* Were receiving welfare benefits in Baltimore, MD
* Received a score of less than or equal to 80% correct on a reading assessment

Exclusion Criteria

* Being at imminent risk for suicide
* Reported hallucinations
* Being incarcerated or otherwise under constant monitoring
* Earned less than or equal to $200 in unreported taxable income from legal activity in the previous month
* Having physical limitations that prevented typing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The results were published in a peer-reviewed journal.

REFERENCES:
- [Result] DeFulio A, Donlin WD, Wong CJ, Silverman K. Employment-based abstinence reinforcement as a maintenance intervention for the treatment of cocaine dependence: a randomized controlled trial. Addiction. 2009 Sep;104(9):1530-8. doi: 10.1111/j.1360-0443.2009.02657.x. PMID 19686522
- [Derived] DeFulio A, Silverman K. Employment-based abstinence reinforcement as a maintenance intervention for the treatment of cocaine dependence: post-intervention outcomes. Addiction. 2011 May;106(5):960-7. doi: 10.1111/j.1360-0443.2011.03364.x. Epub 2011 Mar 7. PMID 21226886

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (N=128) were enrolled in Phase 1 of the therapeutic workplace. Participants (N=51) who became abstinent and skilled were randomly assigned to an Abstinence & Employment (Contingency Management), or an Employment Only group.
Period: Overall Study
Arm/Group | Employment Only | Contingency Management
Started | 24 | 27
Completed | 24 | 26
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Employment Only | Contingency Management | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (7.7) | 43.2 (7.2) | 42.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Monthly Urine Samples That Are Negative for Cocaine
Description: The percentage of urine samples collected at monthly assessments that are negative for cocaine.
Time Frame: 1 year
Measure: Mean (Full Range); unit: percentage of urine samples
Arm/Group | Employment Only | Contingency Management
Number analyzed (Participants) | 24 | 26
percentage of urine samples | 51.8 [0 to 100] | 79.3 [8 to 100]
Statistical Analysis 1: Comparison: Employment Only vs Contingency Management; Test type: Superiority; p = .004, General Estimating Equation (GEE); Odds Ratio (OR) = 3.73, 95% CI 2-sided [1.60 to 8.69]

2. Secondary Outcome: Percentage of Monday, Wednesday and Friday Urine Samples That Are Negative for Cocaine
Description: (The number of Monday, Wednesday and Friday urine samples negative for cocaine/total number of urine samples) x 100.
  We have not confirmed the accuracy/completeness of the Mon, Wed, Fri urine data at this point. In addition, the monthly data had less missing data than the Monday, Wednesday and Friday data and were sufficient to show the main results of the trial.
Time Frame: 1 year
Population: This measure was not analyzed due to limited funding to confirm the accuracy/completeness of the Mon, Wed, Fri urine data
Arm/Group | Employment Only | Contingency Management
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of 30-day Assessment Urine Samples Negative for Opiates
Description: (The number of monthly urine samples negative for opiates/total number of urine samples) x 100
Time Frame: 1 year
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of opiate negative
Arm/Group | Employment Only | Contingency Management
Number analyzed (Participants) | 24 | 27
percentage of opiate negative | 90.6 [25 to 100] | 88.6 [8 to 100]
Statistical Analysis 1: Comparison: Employment Only vs Contingency Management; Test type: Superiority; p = 0.57, General Estimating Equation (GEE); Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.26 to 2.43]

4. Secondary Outcome: Percentage of Monday, Wednesday and Friday Urine Samples That Are Negative for Opiates
Description: (The number of Monday, Wednesday and Friday urine samples negative for opiates/total number of urine samples) x 100.
  We have not confirmed the accuracy/completeness of the Mon, Wed, Fri urine data at this point. In addition, the monthly data had less missing data than the Monday, Wednesday and Friday data and were sufficient to show the main results of the trial.
Time Frame: 1 year
Population: as for outcome 2
Arm/Group | Employment Only | Contingency Management
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: HIV Risk Behaviors
Description: Percentage of people reporting that they traded sex for drugs or money
Time Frame: 1 year
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of participants
Groups:
- Employment Only: Employment Only participants were offered employment for one year, but these participants did not have to provide drug-free urine samples to work.
- Contingency Management: Participants in the Contingency Management group were employed for one year in a Therapeutic Workplace business and had to provide drug-free urine samples to work and earn salary.
Arm/Group | Employment Only | Contingency Management
Number analyzed (Participants) | 24 | 27
percentage of participants | 16.7 [0 to 100] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Employment Only vs Contingency Management; Test type: Superiority; p = 0.046, General Estimating Equation (GEE); Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 0] — The Odds Ratio and Confidence Intervals could not be calculated because one of the groups was at 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Employment Only | Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/27
Serious Adverse Events (participants affected / at risk) | 10/24 | 10/27
Other Adverse Events (participants affected / at risk) | 17/24 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Employment Only (N=24) | Contingency Management (N=27)
Hospitalization for abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hospitalization for anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization for car accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hospitalization for chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization for congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization for depression (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalization for food poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization for high blood sugar (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization for infection (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization for methadone withdrawal (General disorders) | 0 (0) | 1 (1)
Hospitalization for outpatient surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Hospitalization for pinched nerve (Nervous system disorders) | 1 (1) | 0 (0)
Hospitalization for pneumonia (General disorders) | 1 (1) | 2 (2)
Hospitalization for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for infection (Infections and infestations) | 0 (0) | 1 (1)
Incarcerated (Social circumstances) | 1 (1) | 0 (0)
Inpatient drug detoxification, self referred (General disorders) | 0 (0) | 1 (1)
Death, cause undetermined (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Employment Only (N=24) | Contingency Management (N=27)
Anxiety attack, not hospitalized (Psychiatric disorders) | 0 (0) | 1 (1)
Arm, wrist, and/or hand pain, not hospitalized (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Assault, not hospitalized (Social circumstances) | 1 (1) | 1 (1)
Asthma attack, not hospitalized (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain, not hospitalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression, not hospitalized (Psychiatric disorders) | 0 (0) | 1 (1)
E.R. for abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
E.R. for animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
E.R. for asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
E.R. for back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
E.R. for broken bone(s) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
E.R. for chest pains (Cardiac disorders) | 1 (1) | 0 (0)
E.R. for depression (Psychiatric disorders) | 0 (0) | 1 (1)
E.R. for gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (4)
E.R. for general medical treatment (General disorders) | 2 (2) | 3 (3)
E.R for head injury (General disorders) | 0 (0) | 1 (1)
E.R. for hypertension (Vascular disorders) | 0 (0) | 2 (2)
E.R. for infection (Infections and infestations) | 1 (1) | 2 (2)
E.R. for methadone withdrawal (General disorders) | 1 (1) | 0 (0)
E.R. for miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
E.R. for nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
E.R. for pneumonia (General disorders) | 1 (1) | 0 (0)
Injury outside of CLH, not hospitalized (Injury, poisoning and procedural complications) | 4 (4) | 4 (5)
Loss of medical benefits (Social circumstances) | 0 (0) | 1 (1)
Methadone withdrawal, not hospitalized (General disorders) | 1 (1) | 0 (0)
Minor injury at CLH (i.e. scraped knee (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Outpatient dental surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Seizure, not hospitalized (Nervous system disorders) | 1 (1) | 0 (0)
Sick, not hospitalized (General disorders) | 1 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Theft (Social circumstances) | 0 (0) | 1 (1)
Threats of physical violence (Social circumstances) | 4 (5) | 7 (7)
Vomiting (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Wrist injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes